CLINICAL TRIAL: NCT00290316
Title: Accuracy of Endoscopic Ultrasound for Detection of Tumors of the Liver - A Prospective Study
Brief Title: Accuracy of Endoscopic Ultrasound for Detection of Tumors of the Liver
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Central Texas Veterans Health Care System (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0002
Record Dates: First submitted 2006-02-10; First posted 2006-02-13 (Estimated); Last update posted 2006-06-07 (Estimated); Status verified 2006-01

CONDITIONS: Hepatocellular Carcinoma; Hepatoma; Cholangiocarcinoma; Liver Metastases
Keywords: Hepatocellular carcinoma; Cholangiocarcinoma; Metastasis; Liver neoplasm
MeSH Terms: conditions — Carcinoma, Hepatocellular; Cholangiocarcinoma; Neoplasm Metastasis; Liver Neoplasms

INTERVENTIONS:
Procedure: Endoscopy ultrasound

SUMMARY:
The diagnostic accuracy of EUS for detection of the liver tumors (primary and metastatic) remains unknown. To compare the accuracy of the EUS and CT scan for detection of the primary and metastatic carcinoma of the liver.

DETAILED DESCRIPTION:
The incidence of hepatocellular carcinoma is increasing in US. The reason for this increase has been attributed to the emergence of hepatitis C. Studies suggest that patients with hepatitis C are at higher risk of developing hepatocellular carcinoma (elevated alpha-fetoprotein) and, therefore should undergo periodic radiological investigation.

The liver is also a common site for metastases for various malignancies. The metastasis to liver profoundly affects the management and prognosis, since these patients have advanced cancer and therefore are not candidates for surgery.

1.1 Current standards of care

For primary liver tumors alpha-fetoprotein, abdominal ultrasound and CT scan of the abdomen are the suggested tests for the screening in patients that are at higher risk of developing this complication. Measurement of serum alpha-fetoprotein (AFP) may be helpful in the diagnosis and management of HCC. AFP is elevated above 20 ng/Ml in more than 70% of patients with HCC. However, AFP elevations from 10-500 ng/Ml and even occasionally to 1000 ng/ml may be seen in patients with a high degree of inflammatory activity such as with chronic viral hepatitis, who do not have HCC (3). The sensitivity, specificity, and positive predictive value of AFP in 3 well performed screening studies for HCC ranged from 39%-64%, 76%-91%, and 9%-32%, respectively (4). Imaging studies play a key role in the diagnosis of HCC since a significant number of cases are missed by AFP. CT scan and magnetic resonance imaging are commonly used tests.

On the basis of studies conducted over last two decades, National Comprehensive Cancer Network (2004) guidelines for the management of cancer recommended CT scan for the evaluation of the liver for metastases (Please refer to appendix III).

Recent studies have shown that CT scan is far from ideal for detection of primary as well as metastases to liver (5,6). A well designed study showed that CT scan missed 32 % of the primary tumors of the liver. A prospective study of 100 patients with colorectal cancer showed that CT scan missed liver metastases in 37% of cases (5). Another prospective controlled study of 135 subjects showed that CT scan failed to detect liver metastases in 49% of patients with various malignancies (6).

1.2 EUS as a possible diagnostic tool for liver tumors EUS is a well-established tool for the diagnosis and/ or staging of the esophageal, gastric and pancreatic cancer. Recent studies have shown a potential role of EUS for the liver imaging (7, 8, and 9).

1.3 Comparison of EUS and CT scan for detection of liver metastases

Studies suggest that EUS may be an attractive alternative to CT scan for detection of the liver metastases, since it can detect lesions that are missed on the CT scan (9). EUS detected metastatic lesions overlooked by conventional, cross-sectional imaging studies in 5 of 222 cases (2.3%) (9). Another study found occult liver metastases in 2.4% of 574 patients with suspected GI or pulmonary malignancies (4). Each patient found to have occult metastases at EUS had staging CT, which raises an issue as to the quality and/or interpretation of those studies.

An additional advantage of EUS is that fine needle aspiration (FNA) can be performed simultaneously and therefore confirmation of malignancy can usually be accomplished in a single procedure whereas CT or US typically require 2 sessions to accomplish these tasks, one for detection and another for FNA.

1.4 Limitation of EUS: Right lobe The limitation of the EUS is that it is not able to examine the right lobe of the liver completely.

1.5 Rationale for the study. The diagnostic accuracy of EUS for detection of the liver tumors (primary and metastatic) remains unknown. There is sufficient evidence to suggest that EUS may be superior to the CT scan for the liver metastases. Studies that have evaluated the role of EUS are limited by small sample size or retrospective design. Therefore, a prospective study with adequate sample size is required to determine the diagnostic accuracy of endoscopy ultrasound.

2.0 Objectives:

2.1 Primary:

To compare the accuracy of the EUS and CT scan for detection of the primary and metastatic carcinoma of the liver.

2.2 Secondary: 2.2.1 Determine the diagnostic yield of fine needle aspiration using EUS (EUS-FNA) in patients with suspected liver metastasis on EUS examination.

2.2.2 Compare the accuracy of the PET scan with EUS for the detection of the liver metastases.

2.2.3 Determine the safety of EUS-FNA in subjects with liver lesions. 2.2.4 Impact of the EUS on the management of the hepatocellular carcinoma 2.2.5 To study characteristic echoendoscopic findings of the primary and secondary liver tumor.

2.3 Hypothesis: 2.3.1 EUS is likely to detect primary tumor and liver metastasis in subjects with normal CT scan.

3.0 Design: This is a prospective study where study group would comprise of consecutive patients with newly diagnosed colon, pancreatic, esophageal, lung, gastric cancer and patient with hepatitis C or B with elevated levels of alpha-fetoprotein or radiological findings suggestive of mass in the liver.

Patients would be selected from gastroenterology clinic, primary care clinic, surgery clinic, sub-specialty clinics (Oncology, Pulmonary) and hepatitis C clinic. These clinics would be informed about the ongoing EUS study and the eligibility criteria's of the study. All patients will be seen in the gastroenterology clinic where a detail description of the EUS-FNA procedure would be provided to them. In addition, patients would be provided consent forms. (Please refer to section 5 for details of the consent process.)

Study population:

Enrollment of participants.

Patients enrolled in the study would undergo -

* Detailed history and physical examination,
* CT-abdomen preferably with contrast, and
* Possible PET scan. PET scan will be performed on patients who do not have evident distant metastasis.
* Intervention allocation: all eligible patients would be encouraged to undergo EUS and EUS-FNA examination.

Intervention:

Description and schedule: All eligible patients would undergo EUS examination of the liver. Any subject with abnormality suspicious for malignancy in liver would undergo FNA.

Follow-up visits description and schedule. After the procedure patient would be referred back to the clinic from which the patient was identified for further management. These patients are usually seen by oncologists, pulmonologists and cardio-thoracic surgeon depending on the stage and the medical condition of the patient.

ELIGIBILITY:
Inclusion Criteria:

Patients with newly diagnosed colon, pancreatic, esophageal, lung, gastric cancer and patient with hepatitis C or B with elevated levels of alpha-fetoprotein or radiological findings suggestive of mass in the liver.

Exclusion Criteria:

* Advanced heart or lung disease that precludes conscious sedation
* Liver failure

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2004-07; Study Completion 2006-01

PRIMARY OUTCOMES:
To compare the accuracy of the EUS and CT scan for detection of the primary and metastatic carcinoma of the liver.

SECONDARY OUTCOMES:
Secondary:
Determine the diagnostic yield of fine needle aspiration using EUS (EUS-FNA) in patients with suspected liver metastasis on EUS examination.
Compare the accuracy of the PET scan with EUS for the detection of the liver metastases.
Determine the safety of EUS-FNA in subjects with liver lesions.
Impact of the EUS on the management of the hepatocellular carcinoma
2.2.5 To study characteristic echoendoscopic findings of the primary and secondary liver tumor.

CONTACTS AND LOCATIONS:
Overall Officials: Pankaj Singh, MD, Principal Investigator — Central Texas Veterans Health Care System
Locations (1):
- Central Texas Veterans health Care System, Temple, Texas, United States

REFERENCES:
- [Derived] Singh P, Mukhopadhyay P, Bhatt B, Patel T, Kiss A, Gupta R, Bhat S, Erickson RA. Endoscopic ultrasound versus CT scan for detection of the metastases to the liver: results of a prospective comparative study. J Clin Gastroenterol. 2009 Apr;43(4):367-73. doi: 10.1097/MCG.0b013e318167b8cc. PMID 18981929
- [Derived] Singh P, Erickson RA, Mukhopadhyay P, Gopal S, Kiss A, Khan A, Ulf Westblom T. EUS for detection of the hepatocellular carcinoma: results of a prospective study. Gastrointest Endosc. 2007 Aug;66(2):265-73. doi: 10.1016/j.gie.2006.10.053. Epub 2007 Jun 1. PMID 17543307